CLINICAL TRIAL: NCT02122497
Title: The Use of Cardiovascular Biomarkers in Abdominal Aortic Surgery: Possibility of Risk Assessment and Stratification
Brief Title: The Use of Cardiovascular Biomarkers in Abdominal Aortic Surgery
Acronym: BIAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prim PD Dr Afshin Assadian (Other)
Collaborators: Wilhelminenspital Vienna (Other)
Responsible Party: Sponsor-Investigator, Prim PD Dr Afshin Assadian, Prim PD Dr, Wilhelminenspital Vienna
Organization: Wilhelminenspital Vienna (Other)
Other Study IDs: BIAS1.0
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Aortic Aneurysm, Abdominal; Arterial Occlusive Diseases
Keywords: abdominal aortic aneurysm; aortic occlusive disease; cardiovascular biomarkers; open surgical repair; endovascular aortic repair
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Arterial Occlusive Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- abdominal aortic aneurysm (AAA) endovascular: endovascular aortic repair
  Interventions: Procedure: abdominal aortic surgery
- abdominal aortic aneurysm (AAA) open: open surgical repair
  Interventions: Procedure: abdominal aortic surgery
- abdominal aortic occlusive disease (AOD): open surgical repair
  Interventions: Procedure: abdominal aortic surgery

INTERVENTIONS:
Procedure: abdominal aortic surgery
  Other Names: Open surgical repair (OR); Endovascular aortic repait (EVAR)

SUMMARY:
The aim of the present study is the evaluation of cardiovascular biomarkers in patients with abdominal aortic aneurysms (AAA) or abdominal aortic occlusive disease AOD) undergoing open (OR) or endovascular aortic repair (EVAR) with regards to short- and long-term outcome.

By blood collection and measurement of the serum biomarkers Copeptin, N-terminal- pro Brain Natriuretic Peptide (NT-proBNP), cardiac Troponin I (cTnI), high sensitive Troponin T (hs-cTnT) and C-reactive Protein (CRP) we expect an improvement of patients stratification by assessment of cardiac stress tolerance. Data gathered may help to simplify the decision whether an open or endovascular approach for abdominal aortic repair (OR and EVAR) should be performed.

Study Hypothesis:

The evaluation of the predictive value of cardiovascular biomarkers (Copeptin, NT-proBNP, hsTnT, cTnI, CRP) improve patient stratification and selection of surgical treatment.

DETAILED DESCRIPTION:
Background:

The prevalence of coronary artery disease (CAD) in patients with aneurysmal or occlusive disease of the aorta is high: more than 50 percent of patients suffering from peripheral arterial occlusive disease (PAOD) or abdominal aortic aneurysm (AAA) do also have coronary artery disease. As a result, cardiovascular disease is the leading cause of morbidity and mortality in patients undergoing aortic surgery.

Identifying patients at increased risk of cardiac complications following major vascular surgery is also part of the decision-finding process when patients are assigned to open or endovascular surgery. The 30-day mortality rate for elective open aneurysm repair (OR) is estimated to be 4 to 8%, while endovascular aneurysm repair (EVAR) has a perioperative risk of 1.2 to 1.6%. However, the early survival advantage of patients undergoing EVAR disappears with time and all-cause mortality is similar for EVAR and open repair at late follow-up. Patients treated by EVAR show a higher number of complications and reinterventions, and a significant proportion of late deaths after EVAR are due to aneurysm rupture.

Therefore, patients who need abdominal aortic surgery are required to undergo a thorough medical examination, on the one hand to assess cardiac capacity, on the other hand to estimate life expectancy. Current recommendations for the preoperative management of patients undergoing major non-cardiac vascular surgery include physical examination and routine performance of electrocardiogram and echocardiogram as part of a cardiovascular evaluation. However, guidelines do not include routine screening with cardiac enzymes or cardiac stress markers.

Biomarkers:

Brain natriuretic peptide (BNP) and the inactive precursor N-terminal prohormone of brain natriuretic peptide (NT-proBNP) are valuable screening tools for identifying patients who may suffer from heart failure. NT-proBNP plays an important role in heart remodeling and volume homeostasis. It is an important indicator of prognosis in heart failure and after acute myocardial infarction. Elevated pre- and postoperative plasma NT-proBNP levels independently predict postoperative myocardial injury, which is associated with adverse outcome in the short- and long-term regardless of the presence of symptoms of acute coronary syndrome.

Copeptin is a novel marker that allows highly sensitive but unspecific assessment of stress. Copeptin is the C-terminal fragment of provasopressin, the precursor peptide of vasopressin (antidiuretic hormone). Vasopressin is released by the neurohypophysis in order to promote water absorption and vasoconstriction, and thereby contributes to osmotic and cardiovascular homeostasis. Due to the fact that Vasopressin is unstable in the peripheral circulation, the stable Copeptin, which is released in equimolar amounts, is measured instead of Vasopressin. Recent studies have shown that this peptide may also be applied for the assessment of the risk of morbidity and mortality: increased copeptin levels are associated with poor short- and long- term prognosis after myocardial infarction and stroke.

Troponins are widely used biomarkers for the diagnosis and management of acute myocardial infarction and acute coronary syndrome. Troponin is an essential protein of muscle cells. Thus, damage to the heart muscle, such as coronary vasospasm, cardiomyopathy, heart failure and myocarditis, can be indicated by elevated serum levels of cardiac troponin. The most common cause of raised troponins is myocardial ischemia as a result of acute coronary syndrome or myocardial infarction. In patients undergoing major vascular surgery even early small postoperative rises in troponin have been shown to correlate with adverse short- and medium-term outcome.

C-reactive protein (CRP), an acute-phase protein, is a sensitive marker of inflammation and tissue damage. Elevated CRP levels are able to predict future atherothrombotic events, such as stroke, coronary events and progression of peripheral arterial disease. Furthermore, inflammation is crucially involved in atherosclerosis and plaque development.

Material and Methods:

Study Design Prospective, non-randomized, open-labeled, observational study

Patient Population:

500 patients of the Department of Vascular and Endovascular Surgery of the Wilhelminenhospital (Vienna). Preoperative evaluation includes electrocardiography, echocardiography and internal medical examination. Comorbidities, history of cardiac events, previous operations, routine laboratory tests and current medication are documented.

Blood Sampling and Laboratory Measurements:

Blood samples are obtained by venipuncture and collected in standard serum and EDTA tubes preoperatively, 48 hours postoperatively, ten days and six weeks after surgery, centrifuged for 20 minutes at 2000 G and the plasma is stored in aliquots at minus 80 degrees Celsius until determination of the respective biomarkers.

Surgical procedures:

Surgery is standardized by performing endovascular aortic repair (EVAR) or open surgical procedures (OR). OR is performed in general anesthesia via a transabdominal or retroperitoneal approach that allows repair of the aneurysmal or stenosed aorta with tube- or bifurcated grafts. In contrast, groin access for EVAR is achieved in local anesthesia.

Statistical Analysis:

The study cohort consists of three study groups: patients with AAA undergoing EVAR, patients with AAA undergoing OR and patients suffering from AOD undergoing open surgical repair. All patients will be observed until complete follow-up (plasma samples at 0, 2 days, 10 days, 6 weeks and an annual outpatient checkup thereafter) or until a primary fatal outcome event. The statistical distribution of the serum levels of the respective biomarkers is assessed by a histogram. The skewed distribution prompts non-parametric tests (Mann-Whitney-U) for comparison of medians by (gender and status of survival). The effect of biomarkers on 5-year postoperative survival (primary endpoint) is estimated in uni- and multivariate proportional hazard models (Cox Regression) for establishment of a prognostic model. In order to adjust for confounders, the latter includes classic cardiovascular risk factors (age, hypertension, nicotine abuse, diabetes mellitus, history of cardiac events, high lipoproteins), which are documented preoperatively and entered as covariates. Survival estimates stratified by the three study groups will be shown in Kaplan Meier Curves (log-rank test). A two-sided p-value (P) of less than 0.05 is considered to indicate statistical significance. Hosmer and Lemeshow tests are performed to test for adequacy for all regression models (P > 0.05). Tests for proportional hazard assumption is performed through linear regression of partial residuals (Schoenfeld) for each variable and 5-year survival time. Cox proportional hazards model are presented as hazard ratio (HR) and 95% confidence interval (CI). All statistical analyses are performed with the use of SPSS 20 (IBM Inc., Somers, NY 10589, USA.).

ELIGIBILITY:
Inclusion Criteria:

* abdominal aortic aneurysm
* peripheral aortic occlusive disease
* age > 18 years
* approval to participate

Exclusion Criteria:

* absence of clearing for surgery
* canceled surgery
* unability or refusal to participate
* lack of complete follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from abdominal aortic aneurysm or abdominal aortic occlusive disease scheduled either for open surgical repair or endovascular procedure
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
cardiovascular morbidity and mortality | up to five years

SECONDARY OUTCOMES:
all cause mortality | up to five years

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Assadian, PD Dr., Principal Investigator — Department of Vascular and Endovascular Surgery, Wilhelminenhospital Vienna
Locations (1):
- Department of Vascular and Endovascular Surgery, Wilhelminenhospital, Vienna, Vienna, Austria